CLINICAL TRIAL: NCT00886483
Title: Pilot Explorations of Neurofeedback Issues in ADHD
Brief Title: Pilot Feasibility Study of Neurofeedback for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L. Eugene Arnold (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Brain Resource Center (Other)
Responsible Party: Sponsor-Investigator, L. Eugene Arnold, Professor Emeritus, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008H0019-A; 1R34MH080775-01A1 (NIH)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Neurofeedback
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active neurofeedback (Active Comparator): In the active neurofeedback condition, the intervention is active neurofeedback (actual neurofeedback) either twice weekly or three times a week (randomized to frequency), with the same amount of total treatment over 40 sessions, varying only in frequency. Neurofeedback will be via the CyberLearning technology, using videogame race car speed and steering as feedback governed by EEG theta-beta ratio through the interface. the game controller is used in the usual fashion, but maximal speed is capped by the threshold theta-beta ratio, which changes from minute-to-minute by fuzzy logic based on the previous minute's ratio. If theta power exceeds a threshold, the rumble function of the controller comes on as a warning. The feedback is transparent to the patient, who just plays the videogame.
  Interventions: Device: Active Neurofeedback
- Sham Neurofeedback (Sham Comparator): The sham condition will appear identical to the neurofeedback in all aspects: equipment, duration, frequency, and videogame choices. The only difference is that the interface module will be pre-programmed to give random feedback rather than contingent on the participant's brainwave power spectrum.
  Interventions: Device: Sham neurofeedback

INTERVENTIONS:
Device: Active Neurofeedback — A comparison of active neurofeedback to sham neurofeedback and of two treatment schedules: twice weekly vs. three times a week, with the same amount of total treatment over 40 sessions, varying only in frequency.
  Other Names: Electroencephalographic biofeedback, EEG biofeedback
  Arms: Active neurofeedback
Device: Sham neurofeedback — Active neurofeedback vs. sham neurofeedback for 40 treatments, either twice or three times per week.
  Other Names: Electroencephalographic biofeedback or EEG biofeedback
  Arms: Sham Neurofeedback

SUMMARY:
Neurofeedback is increasingly advocated for treatment of ADHD despite a thin evidence base. The numerous open and partially controlled studies suffer serious design flaws. In particular, there is no published double-blind randomized clinical trial (RCT), which would control for experimenter and participant biases. The primary aim of this R34 pilot study is to conduct a small-scale pilot with 39 8-12 year-olds with ADHD to prepare for such a larger RCT.

DETAILED DESCRIPTION:
Thirty-nine boys and girls aged 6-12 with rigorously diagnosed DSM-IV ADHD not currently taking medication will be twice-randomized: first to active neurofeedback (n=26) vs. sham neurofeedback (n=13), and simultaneously to 2 vs. 3 times a week treatment frequency (at least 18 in each frequency, 12 active and 6 sham) for 40 treatments. At treatment 24, major assessments will include measures of satisfaction and blinding, and subjects will be given the option of switching to the opposite treatment frequency for the remaining 16 treatments to generate a practical measure of schedule palatability. Major assessments (at baseline, treatment 12, treatment 24, treatment 40, and follow-up) will include measures of symptoms, functional impairment, academic performance/achievement, and neuropsychological tests of attention, vigilance, and executive functioning. Every 3 treatments parents will rate ADHD symptoms and every 6 treatments teachers will rate, to track the response curve over time. Baseline EEG arousal and ADHD subtype will be examined as possible moderators. By determining the optimal frequency and number of treatments and demonstrating feasibility of double blinding, this pilot study should pave the way for a definitive large RCT of neurofeedback.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 inclusive.
* Boys and girls.
* Primary diagnosis of ADHD, inattentive or combined type.
* Not currently taking medication for ADHD.
* Primary caretaker who can provide frequent parent ratings.
* Item mean ≥1.5 on a 0-3 metric on parent/teacher ratings of DSM-IV inattentive symptoms or on parent/teacher ratings of all 18 ADHD symptoms (while off medication).
* IQ 80 or above and mental age of 6 years or more.
* Willingness and ability to come for 40 treatment sessions and to cooperate with assessments.
* Informed consent and assent

Exclusion Criteria:

* Comorbid disorder requiring psychoactive medication including psychosis, bipolar disorder, severe major depression, and severe anxiety disorders. Patients with mild depression or anxiety not requiring pharmacotherapy will be included and the comorbid symptoms will be tracked.Pervasive developmental disorder is exclusionary by DSM-IV definition of ADHD.
* Medical disorder requiring systemic chronic medication that has confounding psychoactive effects. Asthma inhalants will be allowed, but not chronic systemic corticoids.
* Mental Retardation.
* Anything that would interfere with assessments or study treatment or contraindicate study treatment.
* Plans to move requiring school change during the next 4 months.
* Antipsychotic agent in the 6 months prior to baseline assessment, fluoxetine or atomoxetine in the 4 weeks prior to baseline, stimulant in the week prior to baseline, or other psychiatric medication in the two weeks prior to baseline.
* Previous neurofeedback training of more than 5 treatments.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Eugene Arnold, M.Ed., M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Nisonger Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Lofthouse N, Arnold LE, Hersch S, Hurt E, DeBeus R. A review of neurofeedback treatment for pediatric ADHD. J Atten Disord. 2012 Jul;16(5):351-72. doi: 10.1177/1087054711427530. Epub 2011 Nov 16. PMID 22090396
- [Result] Arnold LE, Lofthouse N, Hersch S, Pan X, Hurt E, Bates B, Kassouf K, Moone S, Grantier C. EEG neurofeedback for ADHD: double-blind sham-controlled randomized pilot feasibility trial. J Atten Disord. 2013 Jul;17(5):410-9. doi: 10.1177/1087054712446173. Epub 2012 May 22. PMID 22617866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: August 2008 to December 2009. Location: Nisonger Center, OSU Medical Center
Pre-assignment Details: Exclusion criteria: IQ <80, mental age <6, comorbid disorder or a medical disorder requiring medication that had psychoactive effects, >5 previous NF treatments, antipsychotic medication within 6 mths pre-baseline, fluoxetine/atomoxetine 4-wks pre-baseline, stimulant 1-wk pre-baseline, or any other psychotropic medication 2-wks pre-baseline.
Groups:
- Active Neurofeedback: In the active neurofeedback condition, subjects will receive accurate neurofeedback either twice weekly vs. three times a week, with the same amount of total treatment over 40 sessions, varying only in frequency.
Period: Overall Study
Arm/Group | Active Neurofeedback | Sham Neurofeedback
Started | 26 | 13
Completed 20 Treatments | 25 | 11
Completed | 24 | 10
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pursue medications | 1 | 2
Not completed — Distance to center, poor grades | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Neurofeedback | Sham Neurofeedback | Total
Number analyzed (Participants) | 26 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 13 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.5) | 8.7 (2.1) | 8.9 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 22 | 4 | 26
Region of Enrollment [Number; unit: participants]
  United States | 26 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Double-blind, Sham-controlled Design #1. Recruitment Number
Description: The feasibility of the double-blind, sham-controlled design was examined in 3 ways, this first way was via the number of participants recruited.
Time Frame: 2 years
Population: Based on inclusion & exclusion criteria and randomization in a 2:1 ratio to active NF vs. sham NF.
Measure: Number; unit: participants
Groups:
- Neurofeedback: In the active neurofeedback condition, subjects will receive accurate neurofeedback either twice weekly vs. three times a week, with the same amount of total treatment over 40 sessions, varying only in frequency.
Arm/Group | Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 26 | 13
participants | 26 | 13

2. Primary Outcome: Feasibility of Double-blind, Sham-controlled Design #2. Retention
Description: The feasibility of the double-blind, sham-controlled design was examined in 3 ways. The second way was via the percentage of participants retained the end of treatment (40th session).
Time Frame: 40th treatment sessions ~ 13-20 weeks
Population: Number randomized was denominator for percentage of participants completing 40 treatment sessions.
Measure: Number; unit: percentage of participants
Groups:
- Active Neurofeedback: Number of participants in the Neurofeedback group (n=26) that completed treatment through the 40th treatment (n=24).
- Sham Neurofeedback: Number of participants in the Sham Neurofeedback group (n=13) that completed treatment through the 40th treatment (n=10).
Arm/Group | Active Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 26 | 13
percentage of participants | 92.3 | 76.9

3. Primary Outcome: Feasibility of Double-blind, Sham-controlled Design #3. Validity of Blind
Description: The feasibility of the double-blind, sham-controlled design was examined in 3 ways. The 3rd way was the percentage of child and parent post-hoc guess regarding treatment assignment.
Time Frame: Post-treatment at session 40
Population: Participants in both Active and Sham Neurofeedback completing 40 treatment sessions.
Measure: Number; unit: percentage of participants
Groups:
- Active Neurofeedback: Correct guess vs. incorrect guess/don't know/decline to guess for Neurofeedback group.
- Sham Neurofeedback: Correct guess vs. incorrect guess/don't know/decline to guess for Sham Neurofeedback group.
Arm/Group | Active Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 24 | 10
percentage of participants
  Declined to guess by children | 35 | 35
  Declined to guess by parent | 29 | 29
  Correct guesses by children | 32 | 32
  Correct guesses by parents | 24 | 24
  Incorrect guesses by children | 32 | 32
  Incorrect guesses by parent | 47 | 47

4. Primary Outcome: Frequency Advisability Outcome (2X vs. 3X/wk) #1 Parent & Child Satisfaction
Description: Parent & child satisfaction of treatment frequency (x2 vs x3 treatments per week) was measured on a likert scale with anchors 0 (indicating low satisfaction) and 7 (indicating high satisfaction).
Time Frame: 24 treatments ~ 8-12 weeks
Population: Those completing 24 treatments
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Neurofeedback: Number of participants in the Neurofeedback group (n=26) that completed treatment through the 24th treatment (n=24).
- Sham Neurofeedback: Number of participants in the Sham Neurofeedback group (n=13) that completed treatment through the 24th treatment (n=10).
Arm/Group | Active Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 24 | 10
units on a scale
  x2 wk Satisfaction | 5.21 (1.80) | 5.40 (1.07)
  x 3/wk Satisfaction | 5.62 (1.27) | 5.08 (1.73)

5. Primary Outcome: Frequency Advisability Outcome (2X vs. 3X/wk) #2. Treatment Frequency Choice
Description: Treatment frequency preference when given choice to change or not to change treatment frequency from 2 to 3X/wk or 3 to 2X/wk at treatment # 24.
Time Frame: 24 treatments ~ 8-12 weeks
Population: participants completing treatment 24
Measure: Number; unit: percentage of participants
Arm/Group | Active Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 24 | 10
percentage of participants
  % participants changing from x2-3 treatments/week | 44 | 44
  % participants changing from x3-2 treatments/week | 22 | 22

6. Primary Outcome: Necessary Duration of Treatment
Description: The necessary duration of treatments was examined via identifying the number of treatments at which improvement stabilized, as shown visually on graphs of parent-rated ADHD symptoms from the SNAP-IV (0-3 scale, lower score is better) for those participants in the Active Neurofeedback who completed 40 treatment sessions.The Sham group is not included in this outcome.
Time Frame: 40 treatment sessions ~ 13-20 weeks
Population: Number of participants in active (n=24) and sham (n=10) neurofeedback completing 40 treatments.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Neurofeedback: All participants in the Active group completing 40 treatments
- Sham Neurofeedback: Participants in the Sham group completing 40 treatments
Arm/Group | Active Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 24 | 10
units on a scale
  SNAP-IV Score Total at Baseline | 1.91 (0.51) | 1.86 (0.44)
  SNAP-IV Score Total at Treatment 12 | 1.52 (0.63) | 1.51 (0.46)
  SNAP-IV Score Total at Treatment 24 | 1.48 (0.60) | 1.56 (0.52)
  SNAP-IV Score Total at Treatment 40 | 1.56 (0.70) | 1.42 (0.58)

ADVERSE EVENTS:
Time Frame: 40 treatment sessions
Arm/Group | Active Neurofeedback | Sham Neurofeedback
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/13
Other Adverse Events (participants affected / at risk) | 0/26 | 0/13

LIMITATIONS AND CAVEATS:
1. Small sample.
2. Self-selection families willing to stop/delay meds.
3. Failure to select for high TBR.
4. Small/medium pre-post ES suggests particular Tx technology may not have been the most effective.
5. Sham NF may not have been inert.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No